CLINICAL TRIAL: NCT06808763
Title: Effect of an Exercise Program on Knee Joint Rehabilitation in Football Players with Anterior Cruciate Ligament Injuries: an Experimental Trial
Brief Title: Exercise Program for Knee Recovery in Football Players with ACL Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Norah A. Alshehri, Consultant and associate professor, King Saud University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RSPD-2025R1090
Record Dates: First submitted 2025-01-21; First posted 2025-02-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: ACL Injuries
Keywords: Anterior Cruciate Ligament (ACL) Injury; Knee Rehabilitation; Muscle Strength; Range of Motion
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rehabilitation Exercise Program for ACL Injury (Experimental): This arm includes a structured rehabilitation exercise program designed to improve knee function, muscle strength, and range of motion in football players with anterior cruciate ligament (ACL) injuries.
  The program is conducted over 22 weeks. Measurements of thigh and leg muscle strength, as well as knee range of motion, are taken at baseline, midway, and post-intervention to evaluate the program's effectiveness.
  This arm aims to assess whether the exercise program restores knee function and supports a safe return to sports.
  Interventions: Other: Knee Rehabilitation Exercise Program

INTERVENTIONS:
Other: Knee Rehabilitation Exercise Program — Rehabilitation Program Description:
  The rehabilitation program was designed to restore knee function and strength progressively in football players recovering from anterior cruciate ligament (ACL) injuries. Key elements of the program are detailed below:
  Program Components:
  Session Structure:
  Each session lasted 60 to 90 minutes. Sessions were performed multiple times weekly, progressively adjusted throughout the program.
  Session Breakdown:
  Warm-Up and Jump Exercises (Part 1):
  Focused on preparing the body for physical activity and improving jump dynamics.
  Dynamic Exercises (Part 2):
  Included drop-jumps, side-hops, and crossover-hops for dynamic knee stabilization and balance.
  Strength Exercises:
  Targeted muscle groups included hamstrings, quadriceps, and calves. Exercises consisted of one-legged leg press, eccentric leg press, squats, one-legged squats on a balance mat, one-legged leg curls, Nordic hamstring, one-legged toe-raises, and lunge exercises.
  Resistance training was i

SUMMARY:
This study aims to evaluate the effectiveness of a structured exercise program in improving knee function, muscle strength, and range of motion in football players recovering from anterior cruciate ligament (ACL) injuries. The study seeks to answer whether a rehabilitation program can restore the performance of the injured leg to levels comparable to the uninjured leg and significantly improve knee functionality over time.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injuries are among the most common and challenging injuries faced by athletes, particularly football players. These injuries can significantly impact knee stability, muscle strength, and range of motion, making effective rehabilitation essential for a full recovery and return to sports.

This study investigates the impact of a structured exercise program on knee rehabilitation in male football players aged 18-22 years with ACL injuries. The goal is to understand whether this program can restore knee function and strength in the injured leg to levels comparable to the uninjured leg.

The rehabilitation program is designed to be implemented over 22 weeks, starting with five sessions per week and tapering to three sessions per week in the later stages. The program focuses on progressively strengthening the thigh and leg muscles, improving knee flexibility, and enhancing overall joint function.

The study uses a pre- and post-measurement experimental design with a single group of participants. The results will help determine whether structured exercise programs can effectively rehabilitate the knee after ACL injuries, enabling football players to regain performance and reduce the risk of future knee problems.

The findings will contribute valuable insights for sports medicine professionals, physiotherapists, and trainers in developing evidence-based rehabilitation protocols for athletes.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed injury to the Anterior Cruciate Ligament (ACL).
* Currently active in playing football.

Exclusion Criteria:

* History of previous surgery to the knee.
* Presence of other musculoskeletal injuries.
* Diagnosis of chronic health conditions.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Outcome Measure: Muscle Strength of the Injured Leg | 22 weeks
  Outcome Measure: Muscle Strength of the Injured Leg Description: Improvement in muscle strength of the injured leg, specifically targeting hamstrings and quadriceps.
  Method of Measurement: Measured using an isokinetic dynamometer at 60°/second angular velocity.
  Unit of Measure: Peak torque (Newton-meters, Nm).

SECONDARY OUTCOMES:
Comparison of Injured and Uninjured Leg Strength | 22 weeks
  Outcome Measure: Comparison of Injured and Uninjured Leg Strength
  * Description: Change in the strength discrepancy between the injured and uninjured legs.
  * Method of Measurement: Measured via isokinetic testing.
  * Unit of Measure: Percentage difference in peak torque between the legs.
  * Time Frame: Baseline, mid-program (11 weeks), and post-program (22 weeks).

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) collected in this study due to data privacy regulations, ethical considerations, and institutional policies.